CLINICAL TRIAL: NCT04927572
Title: A Phase I/IIa Randomized, Double-Blind, Vehicle-Controlled Clinical Trial With Separate Open-Label Active Treatment Phase Evaluating the Safety, Pharmacokinetics and Efficacy of FMX114 Gel in the Treatment of Mild-to-Moderate Atopic Dermatitis in Adults
Brief Title: Safety, Pharmacokinetics and Efficacy of FMX114 Versus Vehicle in Adults With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VY2021-01
Record Dates: First submitted 2021-06-02; First posted 2021-06-16 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMX114 (Experimental)
  Interventions: Drug: FMX114
- Vehicle (Placebo Comparator)
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: FMX114 — Active Comparator
  Arms: FMX114
Other: Vehicle — Placebo Comparator
  Arms: Vehicle

SUMMARY:
A Phase I/IIa Randomized, Double-Blind, Vehicle-Controlled Clinical Trial with Separate Open-Label Active Treatment Phase Evaluating the Safety, Pharmacokinetics and Efficacy of FMX114 Gel in the Treatment of Mild-to-Moderate Atopic Dermatitis in Adults

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have the ability to understand and be willing to sign an informed consent form.
2. Aged ≥ 18 years, at time of screening visit.
3. Weight ≥ 40 kg, at time of screening visit.
4. Diagnosis of Atopic Dermatitix with a total body surface area (BSA) of AD involvement of ≤ 35% excluding involvement of face, scalp and groin at screening and Day 1, prior to first dose.
5. Atopic dermatitis should be present for at least 3 months with stable disease for ≥ 1 month at the time of the screening visit and on Day 1, prior to dose administration.
6. Have the presence of at least 2 comparable target AD lesions (size approximately 10 to 200 cm2), located on the trunk, upper extremities or lower extremities. In addition, the 2 target lesions:

   1. must have ADSI score of ≥ 6 and ≤ 12 AND a between-lesion difference in ADSI of ≤ 1.
   2. must be separated by ≥ 10 cm.
7. Positive varicella zoster virus (VZV) antibody test at the screening visit. At the discretion of the Investigator, subjects who return a negative result may be re-screened following a full VZV vaccination course.
8. Medically healthy in the opinion of the Investigator without significant abnormalities at the screening visit and prior to dose administration on Day 1, including:

   1. Physical examination without any clinically relevant findings (excluding findings relating to AD).
   2. Systolic blood pressure in the range of 90 to 160 mmHg (inclusive) and diastolic blood pressure in the range of 50 to 95 mmHg (inclusive) after 5 minutes in supine position.
   3. Heart rate in the range of 45 to 100 bpm (inclusive) after 5 minutes rest in supine.
   4. Body temperature (tympanic or oral), between 35.5°C and 37.7°C (inclusive).
   5. Electrocardiogram findings (ventricular HR, PR interval, QRS duration, QT interval and QTcF) within normal ranges (site-specific normal ranges may be used).
   6. Triplicate 12-lead electrocardiogram (ECG) (taken after the subject has been supine for at least 5 minutes) with a QTcF ≤ 450 msec for males and ≤ 470 msec for females and no other clinically significant abnormalities.
   7. All laboratory blood and urinalysis test results within normal ranges for the local laboratory, including the following specific findings:

   i. Lymphocyte count ≥ 0.5 x 10 9/L ii. Haemoglobin ≥ 9g/dL iii. Absolute neutrophil count ≥ 1 x 10 9/L Assessments may be repeated once, if abnormal values were recorded in the first instance, at the discretion of the PI.
9. Female subjects must:

   * Be of non-childbearing potential (i.e., surgically sterilised [hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 weeks before the screening visit]) or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause, and a follicle-stimulating hormone [FSH] level >40 IU/L at the screening visit), or
   * If of childbearing potential, must agree not to donate ova, not to attempt to become pregnant and, if engaging in sexual intercourse with a male partner, must agree to use an acceptable method of contraception (refer to Section 21.5) from signing the consent form until at least 2 months after the last dose of the study drug.
10. Male subjects, if not biologically or surgically sterilized, must agree not to donate sperm and, if engaging in sexual intercourse, must agree to use a condom from signing the consent form until at least 90 days after the last dose of study drug. If engaging with a female partner who could become pregnant, the female partner must additionally use an acceptable method of contraception (refer to Section 21.5) for this same period.
11. Have suitable venous access for blood sampling.
12. Be willing and able to comply with all study assessments (optional photography assessments excluded) and adhere to the protocol schedule and restrictions

Exclusion Criteria:

1. In the opinion of the Investigator, subject has unstable or actively infected AD at the screening visit, or prior to dose administration on Day 1.
2. Active impetigo at any of the target lesions.
3. Concomitant dermatologic conditions (e.g. irritant contact dermatitis, allergic contact dermatitis, psoriasis, etc.) or other medical condition(s) which may, in the opinion of the Investigator, interfere with evaluations of the subject's response to study drug.
4. Positive test results for active human immunodeficiency virus (HIV-1 or HIV-2), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
5. Evidence or history of active, latent or inadequately treated tuberculosis (TB) infection at the screening visit.
6. Evidence or history of disseminated or recurrent herpes zoster infection.
7. Clinically significant active infection (in the opinion of the Investigator) within 2 weeks prior to first dose application on Day 1.
8. Any known or suspected premalignant or malignant disease within the last 5 years (excluding successfully treated basal cell carcinomas).
9. Have received AD-directed therapy within the following timeframes prior to dose administration on Day 1:

   1. Ultraviolet A (UVA) or Ultraviolet B (UVB) therapy within 2 weeks.
   2. Systemic or topical corticosteroids within the past 2 weeks.
   3. Other topical anti-inflammatory therapy e.g. Janus kinase (JAK) inhibitors, calcineurin inhibitors, Phosphodiesterase-4 inhibitors within the past 2 weeks.
   4. Systemic JAK inhibitors within the past 12 weeks.
   5. Systemic biologic therapy within the past 12 weeks.
   6. Bleach or other antiseptic baths (e.g., potassium permanganate) within the past 2 weeks.
   7. Any other active topical therapy on target lesions within 7 days (does not include non-medicated moisturisers, sunscreens, lotions or creams).
10. Use of any topical product (e.g. sunscreen, lotions, creams) on the target lesion within 24 hours prior to dose administration on Day 1.
11. Live and live attenuated vaccines are not permitted within 30 days prior to the first application of study drug, and for 2 months following the last dose application. It is noted that mRNA or adeno-associated virus (AAV)-based COVID-19 vaccinations are permitted at any stage throughout the study.
12. Use of any systemically absorbed prescription or over-the-counter medication (including herbal products, diet aids, and hormone supplements) within 10 days or 5 half-lives of the medication (whichever is longer) prior to the first study drug administration Exceptions may be made for medications which, in the opinion of the Investigator, are unlikely to affect the course of the AD during the study period (for example stable use of antihistamines for asthma or allergies. Antibiotics, if not known to impact AD disease course, may also be allowed at the discretion of the PI in consultation with the medical monitor).
13. Participation in another investigational clinical trial within 30 days (or 5 half-lives, of the investigational agent) (whichever is longer) prior to the first study drug administration.
14. Presence or evidence of recent sunburn, scar tissue, tattoo (more than 25% of body area), open sore, or branding that, in the opinion of the Investigator, would interfere with evaluations of the subject's response to study drug.
15. Known hypersensitivity to any component of the study drug.
16. Demonstrated clinically significant (required intervention, e.g., emergency room visit, epinephrine administration) allergic reactions (e.g., food, drug, or atopic reactions, asthmatic episodes) which, in the opinion of the Investigator, would interfere with the subject's ability to participate in the trial.
17. Known or suspected history of alcohol or drug abuse (in the opinion of the Investigator) within the last 2 years.
18. Documented history of depression or self-harm that is not, in the opinion of the Investigator, currently adequately controlled with medication or in remission.
19. Positive drug or alcohol test results at the screening visit or on Day 1, prior to dose administration (may be repeated once, if a positive test was recorded in the first instance, at the discretion of the Investigator).
20. Consumption of grapefruit or Seville orange (or products containing grapefruit or Seville orange) within 72 hours prior to the first FMX114 dose administration on Day 1 (consumption is also not permitted throughout the duration of the study).
21. Any other condition or prior therapy that in the opinion of the Investigator would make the subject unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Atopic Dermatitis Severity Index (ADSI) score at Day 29 | Day 29
Incidence, type and severity of adverse events (AEs) at Day 43 | Day 43

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Investigator #9, Miami, Florida
  - Investigator #14, Miami, Florida
  - Investigator #12, Miramar, Florida
  - Investigator #13, Sugarloaf, Pennsylvania
- Australia (3):
  - Investigator #5, Phillip, Australian Capital Territory
  - Investigator #6, Darlinghurst, New South Wales
  - Investigational Site #1, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No